CLINICAL TRIAL: NCT03691285
Title: Mandibular Overdenture Retained by 1 or 2 Implants: a Cost-effectiveness Analysis
Acronym: IOD1-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, Cláudio Rodrigues Leles, Associate Professor, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI087-2017
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Edentulous Mouth
Keywords: Overdenture; Dental implant; Cost analysis
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Intervention Model Description: Comparative effectiveness of two competing strategies for the edentulous mandible using implants
Masking Description: To avoid selection bias and ensure adequate allocation concealment, their treatment group will only be revealed for each participant after the assessment of the baseline outcomes, which will occur after the delivery and regular use of the new set of conventional dentures. Since full blinding for the two interventions is not possible for those involved with treatment management and collection of data, only those collecting and analyzing clinical data from masticatory performance tests will be unaware of the assigned treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-implant mandibular overdenture (Experimental): Participants allocated to this group will have an implant placed in the mandibular midline and after 3 weeks (healing period - early loading) an attachment system will be tightened and a retention matrix will be incorporated to the mandibular denture.
  Interventions: Procedure: Mandibular Overdenture
- Two-implant mandibular overdenture (Active Comparator): Participants allocated to this group will have two implants placed in the inter-foraminal region after 3 weeks (healing period - early loading) an attachment system will be tightened and a retention matrix will be incorporated to the mandibular denture.
  Interventions: Procedure: Mandibular Overdenture

INTERVENTIONS:
Procedure: Mandibular Overdenture — Placement of 1 or 2 implants in the anterior region of the edentulous mandible.

SUMMARY:
The aim of this study is to assess the cost-effectiveness of the mandibular overdenture retained by one and two implants, based on a randomized clinical trial.

DETAILED DESCRIPTION:
This randomized clinical trial alongside a cost-effectiveness analysis will include 48 edentulous individuals who meet eligibility criteria. New maxillary and mandibular dentures will be fabricated for all participants following a standardized protocol. Then, participants will be randomized into one of the treatment groups: mandibular overdenture retained by two implants group or single-implant mandibular overdenture group. Each participant allocated to the single-implant mandibular overdenture group will then receive a Straumann® Standard Plus SLActive® regular neck implant (Straumann 0.33.051S/052S/053S Institute Straumann AG, Basel, Switzerland) in the mandibular midline, and the mandibular overdenture retained by two implants group will receive two implants of the same specification, in the interphoramen region. A healing abutment will be connected and the implant will be allowed to heal for approximately 3 weeks. Then, a 3.4mm retentive titanium anchor abutment (Straumann 048.439, Institute Straumann AG, Basel, Switzerland) will be connected and tightened to 35 N.cm with a torque wrench. The matrix will be incorporated to the denture using self-curing acrylic resin and the patient will be instructed to keep the upper and lower dentures firmly occluded in the habitual position until the final polymerization of the resin. Outcomes (satisfaction with the dentures and oral health-related quality of life) will be measured at baseline and at the 6- and 12-month follow-up. Direct costs related to therapies in both groups will be identified, measured and valuated for one year after treatment. Incremental cost-effectiveness ratios will be estimated and graphically presented on cost-effectiveness planes. Sensitivity analysis on the most important assumptions will be performed in order to assess the robustness of the model.

ELIGIBILITY:
Inclusion Criteria:

* No contraindications for implant surgery (mainly related to uncontrolled systemic diseases)
* Present enough bone volume in the mandibular midline area for implant placement without the need of bone augmentation procedures.
* Be able to understand and answer the questionnaires used in the study
* Agree to participate by providing a written informed consent.

Exclusion Criteria:

* Noncompliant participants
* Individuals who do not agree to be randomly allocated to the treatment study group
* Presence of signs of untreated temporomandibular disorders, uncontrolled systemic or oral conditions that require additional treatments

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-04-09 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the dentures | Changes from baseline to 12 months after the intervention
  A 100 cm graduated visual analogue scale will be used in order to assess the participants' ratings of their satisfaction with the upper and lower dentures in relation to the parameters "general satisfaction", "comfort", "stability", "aesthetics", "ability to speak" and "ability to chew". Each participant will indicate their level of satisfaction with each parameter by marking a point along the scale, in which ends mean "unsatisfied" and "satisfied", as it is closer to the beginning or the end of the scale, respectively.

SECONDARY OUTCOMES:
Masticatory efficiency | Changes from baseline to 12 months after the intervention
  Masticatory efficiency will be assessed as a secondary outcome using a two-colored chewing gum test and a qualitative and quantitative colourimetric method to measure the color-mixing ability. Participants will be asked to sit upright in a dental chair and to chew the gum on their preferred chewing side for 20 cycles. Visual and electronic analysis of the chewed gums samples will be done according to the classification proposed by Schimmel et al. Analysis will be made by two investigators blinded to the study groups and treatment stage. The software ViewGum (dHAL Software, Kifissia, Greece, www.dhal.com) will be used for electronic colourimetric analysis.
Pain and discomfort | 24 hours, 7 days and 21 days after surgery
  A 100 cm graduated visual analog scale will be used to evaluate participants' assessments of pain and discomfort regarding the surgical process. Each participant will indicate their level of pain and discomfort with each parameter by marking a point along
Oral health-related quality of life impacts | Changes from baseline to 12 months after the intervention
  The cross-culturally adapted Brazilian version of the Oral Health Impact Profile for edentulous subjects (OHIP-EDENT) will be used. It contains 19 items divided in four different subscale domains: (I) masticatory discomfort and disability (four items), (II) psychological discomfort and disability (five items), (III) social disability (five items), and (IV) oral pain and discomfort (five items). The items are answerable by a 3-point Likert scale and responses will be summed to result an overall score. Higher scores represent worse OHRQoL.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry, Federal University of Goias, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: No